CLINICAL TRIAL: NCT03550040
Title: 3D Versus Robot Assisted Laparoscopic Prostatectomy. A Prospective Randomized Non-inferiority Study.
Brief Title: 3D Versus Robot Assisted Laparoscopic Prostatectomy.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: accrual was sufficient at interim analysis to draw final conclusions needed to publish
Sponsor: Tampere University Hospital (Other)
Collaborators: Seinajoki Central Hospital (Other)
Responsible Party: Principal Investigator, Antti Kaipia, Chief physician, department of urology, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18005
Record Dates: First submitted 2018-05-14; First posted 2018-06-08 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: radical prostatectomy; laparoscopic prostatectomy; robot assisted prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot assisted prostatectomy. (Active Comparator): Intervention: radical prostatectomy
  Interventions: Procedure: Radical prostatectomy
- 3D laparoscopic prostatectomy (Experimental): Intervention: radical prostatectomy
  Interventions: Procedure: Radical prostatectomy

INTERVENTIONS:
Procedure: Radical prostatectomy — Surgical removal of the prostate
  Other Names: Total prostatectomy

SUMMARY:
A randomized, prospective study to compare the direct and indirect costs, functional and oncologic results of 3D laparoscopic and robot assisted radical prostatectomy procedures.

DETAILED DESCRIPTION:
The direct and indirect costs, functional and oncologic results of robot assisted radical prostatectomy (RALP) are compared to those of 3D laparoscopic radical prostatectomy. The hypothesis of the study is that the functional and oncologic results of the two operative methods are equal, but the direct costs of RAPL are significantly higher. A randomized, prospective non-inferiority study will will enroll 280 patients randomized 1:1 to both operative approaches to test this hypothesis. The primary functional outcome measure is the proportion of patients with complete urinary continence (no protective pad use) at 12 months post operatively. Secondary functional outcome measure is the preservation erectile function at 12 months post operatively. Oncologic outcome measures are the proportion of patients with undetectable post operative prostate specific antigen levels and positive surgical margins at pathological examination. The direct and indirect costs of both operative approaches are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Localized prostate cancer undergoing radical prostatectomy
* Patient has to understand and be able to write and read Finnish language
* No prior head injury, dementia or Parkinson's disease
* No concomitant malignant illness
* Life expectancy of at least 10 years
* 35-74 years of age

Exclusion Criteria:

* Locally advanced prostate cancer (T4)
* Suspicion or documented metastases (M1)
* Serum PSA > 20 ng/ml
* Prior laparoscopic hernia surgery employing non resorbable mesh
* Prior pelvic irradiation or major surgery
* Prior malignant disease within prior 5 years excluding skin cancer (non-melanoma).

Ages: 34 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Urinary continence | 12 months
  Expanded Prostate Cancer Index Composite (EPIC) Short Form (EPIC-26), urinary domain score is used to assess the return of continence post operatively. The percentage of patients with no protective pad use at 12 months post operatively is the main outcome measure.

SECONDARY OUTCOMES:
Erectile function | 12 months
  International Index of Erectile Function (IIEF-5) Questionnaire score is used to quantify the return of erectile function post operatively.
Prostate specific antigen | 12 months
  Post operative prostate specific antigen levels.
Evaluation of surgical margins at pathologic examination. | up to 12 months
  The oncological outcome is evaluated by the presence of cancerous tissue at the surgical margins of the specimen at pathologic examination.

OTHER OUTCOMES:
costs of treatment | 12 months
  Direct and indirect treatment related costs.

CONTACTS AND LOCATIONS:
Overall Officials: Antti Kaipia, M.D., Ph.D., Principal Investigator — chief, dept of urology
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Yes
Patient demographic, primary and secondary outcome measures available upon request.
Supporting Information: Study Protocol
Time Frame: 2020 onward for 5 years.
Access Criteria: IPD will be made for relevant high quality reseach uopn request.